CLINICAL TRIAL: NCT01683162
Title: Effects of Parenteral Nutrition With Different Lipid Emulsions in Preterm Infants
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wei Cai (Other)
Responsible Party: Sponsor-Investigator, Wei Cai, vice-president, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PNDLEIPI
Record Dates: First submitted 2012-07-18; First posted 2012-09-11 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Preterm Infant
Keywords: parenteral nutrition; lipid emulsion; olive oil; liver function; fatty acid; clinical outcomes
MeSH Terms: conditions — Premature Birth; Hyperphagia | interventions — ClinOleic; Lipofundin; soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Olive oil lipid emulsion (Experimental): the olive oil lipid emulsion is ClinOleic
  Interventions: Drug: ClinOleic
- MCT/LCT lipid emulsion (Experimental): the MCT/LCT lipid emulsion is Lipofundin
  Interventions: Drug: Lipofundin
- LCT lipid emulsion (Experimental): the LCT lipid emulsion is Intralipid
  Interventions: Drug: Intralipid

INTERVENTIONS:
Drug: ClinOleic — the lipid of all-in-one, 0.5-3.5g/kg.d
  Arms: Olive oil lipid emulsion
Drug: Lipofundin — the lipid of all-in-one, 0.5-3.5g/kg.d
  Arms: MCT/LCT lipid emulsion
Drug: Intralipid — the lipid of all-in-one, 0.5-3.5g/kg.d
  Arms: LCT lipid emulsion

SUMMARY:
Previous studies have suggested that olive oil-based emulsion is safe and well tolerated in preterm infants, a showed efficacy and a good clinical and biological safety profile. The objective of this study was to assess the effects of a new olive-oil based lipid emulsion compared with the traditional lipid emulsions.

DETAILED DESCRIPTION:
For a number of years, lipid emulsions have been used in the nutritional support of surgical and critically ill patients, with the aim of supplying substrates to meet energy demands and providing building blocks for wound healing and tissue repair. Two types of lipid emulsions are currently used for adult as well as pediatric patients: one lipid emulsions prepared from soybean oil that are composed of long-chain triacylglycerols (LCTs), 62% of which are polyunsaturated fatty acids (PUFAs), and the other lipid emulsions composed of 50% medium-chain triacylglycerols (MCTs) and 50% LCT soybean oil. A new lipid emulsion prepared from a mixture of soybean oil and olive oil contains only LCTs and has a lower proportion (20%) of PUFAs and 60% monounsaturated fatty acids (MUFAs). There are so many investigations with olive oil-based emulsion including in-vitro studies, animal studies, and infusion studies in healthy subjects and in various patient groups. In-vitro and animal studies demonstrate that the impairment of immune function, especially of T cell responses, that occurs with soybean oil-based emulsions is avoided with ClinOleic. Studies in infants and adults have consistently shown that olive oil-based emulsion increases the oleic acid content of blood lipids and that it avoids the depletion of long chain n-6 PUFA derivatives of linoleic acid that is seen with soybean oil-based emulsion. The less unsaturated nature of olive oil-based emulsion compared will possibly decrease oxidative stress. Further studies are required to test their beneficial effect from olive oil consumption in preterm infants.

The investigators designed a double-blind, randomized clinical trial to performed the effect of lipometabolism, oxidative stress and clinical outcomes of olive oil , MCY/LCT and LCT lipid emulsions.

ELIGIBILITY:
Inclusion Criteria:

* Infants of both genders
* Hospitalized
* The parent of the infant agreed to participate by signing an informed consent form
* Infants admitted hospital within 72 hours after birth(gestational age<37 weeks)
* Birth weight <= 2000g
* No PN support contraindications
* Parenteral nutrition for 14 days or more
* The parent of the infant is to sign an informed consent form prior to enrollment

Exclusion Criteria:

* Receiving PN before screening
* EN caloric>10%
* Obstruction jaundice
* Suspected or identified biliary tract atresia
* Neonatal hepatitis
* Infants with liver markers >2 times normal levels
* Infants with renal markers >2 times normal levels
* Congenital metabolic situations
* Identified as having major chromosomal disease
* CMV, virus hepatitis and syphilis infection
* Congenital or acquired immune deficiency

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2012-07; Primary Completion 2012-12 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
lipometabolism | Change from Baseline in fatty acid at 7 days and 14 days
  fatty acid

SECONDARY OUTCOMES:
oxidative stress | Change from Baseline in liver function at 7 days and 14 days
  superoxidase dismutase(SOD),malondialdehyde(MDA),glutathione peroxidase(GSH-Px),total-anti-oxidizing-capability(T-AOC)

OTHER OUTCOMES:
clinical outcomes | before PN; participants will be followed for the duration of hospital stay, an expected average of 5 weeks
  the growth of weight and head circumference, days on ventilator, length of hospitalization, morbidity of sepsis and NEC

CONTACTS AND LOCATIONS:
Overall Officials: Ying Wang, phd, Principal Investigator — Xin Hua Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai,China
Locations (1):
- Xin Hua Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wang Y, Feng Y, Lu LN, Wang WP, He ZJ, Xie LJ, Hong L, Tang QY, Cai W. The effects of different lipid emulsions on the lipid profile, fatty acid composition, and antioxidant capacity of preterm infants: A double-blind, randomized clinical trial. Clin Nutr. 2016 Oct;35(5):1023-31. doi: 10.1016/j.clnu.2015.10.011. Epub 2015 Oct 31. PMID 26561301